CLINICAL TRIAL: NCT00125502
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled, Clinical Trial of Recombinant CMV gB Vaccine in Postpartum Women
Brief Title: Recombinant CMV gB Vaccine in Postpartum Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Robert Pass, MD (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); MCM Vaccines B.V. (Industry)
Responsible Party: Sponsor-Investigator, Robert Pass, MD, Professor of Pediatrics, University of Alabama at Birmingham
Organization: University of Alabama at Birmingham (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 99-038; U01AI063565 (NIH); sanofi pasteur CMC00
Record Dates: First submitted 2005-07-29; First posted 2005-08-01 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2011-09

CONDITIONS: Cytomegalovirus Infections
Keywords: CMV, Cytomegalovirus, vaccine, women, postpartum
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I (Experimental): n=200; 20 micrograms gB with MF59
  Interventions: Biological: CMV gB vaccine; Drug: MF59 adjuvant
- II (Placebo Comparator): n=200; placebo (normal saline)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: CMV gB vaccine — CMV gB is combined with a novel adjuvant, MF59, a proprietary oil-in-water emulsion, administered at 0, 1, and 6 months.
  Arms: I
Drug: MF59 adjuvant — Oil-in-water emulsion
  Arms: I
Drug: Placebo — Normal saline solution
  Arms: II

SUMMARY:
The purpose of this study is to determine if a new cytomegalovirus (CMV) vaccine (CMV gB/MF59) can safely prevent mothers from catching CMV infection between pregnancies. This study includes 464 women, ages 14-40 years, who delivered a newborn infant within 12 months prior to the study. Participants must live within the Birmingham metropolitan area or the Tuscaloosa county area and they cannot have had CMV infection previously. CMV vaccine or placebo (substance containing no medication) will be given at 3 study visits. Participants fill out diary cards for 7 days after each vaccination. Blood samples will be collected. Urine samples will be collected several times and pregnancy tests will be performed. Participants who tested positive for CMV will have urine, vaginal swab, and saliva specimens collected. Each participant will be followed for 3 years after the third dose of vaccine. Infants born to participants in the study will be checked for CMV infection.

DETAILED DESCRIPTION:
The objective of this double-blind, randomized, placebo-controlled Phase II study is to determine whether a recombinant subunit vaccine comprised of cytomegalovirus (CMV) envelope glycoprotein B (gB) with MF59 adjuvant can prevent maternal CMV infection between pregnancies in a high risk population of women of childbearing age. This study will also permit determination of whether the approach used is a feasible one for a large scale efficacy trial with prevention of congenital CMV as the endpoint. CMV gB vaccine is comprised of a recombinant CMV envelope glycoprotein produced in a Chinese hamster ovary cell line. The CMV gB is combined with a novel adjuvant, MF59, a proprietary oil-in-water emulsion. Vaccines will be administered at 0, 1, and 6 months by intramuscular injection in the left deltoid. Placebo recipients will be given a normal saline solution. Study participants were recruited from postpartum wards and from the community. Potential participants were screened for antibody to CMV; those who were seronegative were invited to participate in the vaccine study. Participants received their initial immunization 1.5 to 12 months postpartum. A total of 464, seronegative women who were willing to participate and met enrollment inclusion and exclusion criteria were randomized to 1 of 2 groups: Group I participants received 20 micrograms of gB with MF59; Group II participants received placebo (normal saline). During the immunization period local and systemic reactogenicity was assessed by a 7-day diary card completed after each dose of vaccine. Adverse events are tabulated. Safety is assessed by comparing the local and systemic reactogenicity and adverse event rates between vaccine and placebo recipients. Study participants are screened for CMV infection every three months, beginning three months after the first dose of vaccine, using a CMV IgG antibody assay with preabsorption of sera with purified recombinant CMV gB (vaccine antigen). CMV infection will be confirmed by either isolation of virus or detection of CMV DNA in body fluids. After the 3 dose vaccine schedule has been completed, participants are followed every 3 months. The primary endpoint is the time to CMV infection. The rate of congenital CMV infection in offspring of immunized mothers is a secondary endpoint. The rate of congenital CMV infection will be compared between offspring of vaccine and placebo recipients. Each subject will be followed for 3 years from the third dose of vaccine. Specific information will be collected on the following pregnancy outcomes: pregnancy report, pregnancy follow-up, abnormal pregnancy outcome-mother, and abnormal pregnancy outcome-infant.

ELIGIBILITY:
Inclusion Criteria:

* Mothers, 14 to 40 years of age (inclusive), who have delivered a newborn infant within the previous 12 months, reside within the Birmingham metropolitan area or the Tuscaloosa county area, and sign an informed consent form following a detailed explanation of the study.
* Cytomegalovirus (CMV) seronegative as determined by the Axsym® System CMV IgG antibody assay (Abbott Diagnostics) performed within 14 weeks prior to the first immunization.
* In good health as judged by medical history obtained by patient interview and physical examination.
* Willing to participate with 4 follow-up visits per year for 3 years after the third dose of vaccine.
* Volunteers must be willing to use an effective means of contraception of their choice from the first dose of vaccine up to 2 months after the third dose of the vaccine.

Methods that were considered effective for the purposes of this clinical trial included any hormonal contraceptive, double barrier methods and abstinence.

Exclusion Criteria:

* Known maternal immune disorder such as HIV infection, collagen vascular disease, immune deficiency, or chronic disease requiring treatment with immunosuppressive medication.
* Chronic disease such as diabetes, sickle cell disease, heart disease, fibromyalgia, arthritis or asthma requiring medication.

Patients with a diagnosis of asthma or past asthma were allowed to enroll if they did not currently take medication for asthma and were off asthma medication and free from asthma symptoms for at least 2 years. Patients with mild to moderate essential hypertension on medication were allowed if their blood pressure was controlled within the normal range for at least one month.

* Positive rapid test for HIV antibody. All subjects were tested for HIV antibody using a rapid serologic test at the time of enrollment beginning with protocol version 1.7. Prior to that only subjects who had a history of a negative screening test for HIV during their most recent pregnancy were included. Subjects given HIV rapid serologic tests in this study were provided pre-test counseling before the test was performed and post-test counseling when the subject was informed of the test results. This counseling is provided by the study nurses according to CDC guidelines [Centers for Disease Control and Prevention. Revised Guidelines for HIV Counseling, Testing and Referral and Revised Recommendations for HIV Screening of Pregnant Women. Subjects who are eligible for this study were considered very unlikely to be HIV positive because almost all adults who are HIV positive are also CMV positive and almost all potential enrollees will have received HIV screening during their recent pregnancy.
* Maternal sterilization procedure planned in the postpartum period.
* Current use of steroids or other immunosuppressive medications.
* Maternal drug or alcohol abuse.
* Mothers who are nursing their infants.
* Participation in a clinical trial of another investigational vaccine or drug, if they have received the investigational drug or vaccine within 6 months prior to enrollment date for this trial.
* A history of anaphylaxis or serious vaccine reactions.
* Previous receipt of CMV vaccine.
* Receipt of blood products within 3 months prior to study enrollment.

Ages: 14 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 464 (Actual)
Dates: Start 1999-08; Primary Completion 2007-06 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Time to CMV infection. | From initial vaccine to final study visit.

SECONDARY OUTCOMES:
Rate of CMV infection in CMV gB vaccine and placebo recipients. | From initial vaccine to final study visit.
Rate of congenital CMV infection in offspring of the immunized women. | From initial vaccine to final study visit.
Rate of local and systemic reactions and adverse events. | Duration of study.
Peak levels of antibody to CMV gB and neutralizing antibody and decline in antibody levels over time. | 2 weeks post third dose of vaccine and decline over time up to 3 years post-third dose of vaccine.
Lymphocyte proliferation response to gB. | From 3 months post-third dose of vaccine to study termination.

CONTACTS AND LOCATIONS:
Overall Officials: Robert F Pass, MD, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Alabama at Tuscaloosa, Tuscaloosa, Alabama

REFERENCES:
- [Derived] Pass RF, Zhang C, Evans A, Simpson T, Andrews W, Huang ML, Corey L, Hill J, Davis E, Flanigan C, Cloud G. Vaccine prevention of maternal cytomegalovirus infection. N Engl J Med. 2009 Mar 19;360(12):1191-9. doi: 10.1056/NEJMoa0804749. PMID 19297572